CLINICAL TRIAL: NCT02655055
Title: Randomized Longitudinal Study of Apheresis Voluntary Blood Donors' Bone Density
Brief Title: Bone Density in Voluntary Apheresis Blood Donors
Acronym: ALTRUYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versiti Blood Health (Other)
Collaborators: Marquette University (Other); Medical College of Wisconsin (Other); University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRO00026241
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Bone Density
Keywords: apheresis; citrate anticoagulation; blood donor; bone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): high frequency voluntary apheresis blood donation (i.e. 20 - 26 donations in one year period)
  Interventions: Procedure: high frequency voluntary apheresis blood donation
- Control (No Intervention): no voluntary (or paid) apheresis blood donation (whole blood donation allowed during one year period)

INTERVENTIONS:
Procedure: high frequency voluntary apheresis blood donation
  Arms: Intervention

SUMMARY:
A longitudinal, randomized, controlled, single-center Phase IV clinical trial will be performed to assess changes in bone mineral density (BMD) among voluntary apheresis blood donors. The primary outcome measure will be clinically significant decline in BMD at the lumbar spine assessed by dual-energy x-ray absorptiometry (DXA).

DETAILED DESCRIPTION:
Apheresis blood donation maximizes an individual's donation by selecting specific blood components that are used to save patient lives. Dramatic increases in the number of apheresis procedures performed each year are apparent both domestically and internationally. Apheresis requires the use of citrate anticoagulation, a substance that confers its anticoagulant effect through chelation of cations, like calcium. A small number of cross-sectional studies have reported that intermittent exposure to citrate through apheresis is associated with significant declines in donor bone mineral density (BMD). In contrast, oral potassium citrate of much lower dose has been used to treat low bone density with well-documented efficacy. The impact of citrate exposure during apheresis, either positive or negative, is important given that BMD is a significant risk factor for low trauma fracture, a problem that affects more than 2M people in the U.S. annually. It is ultimately unknown what effect repeated apheresis has on skeletal health. To address this knowledge gap, we will perform a Phase IV clinical trial of apheresis blood donors using a cross-disciplinary, multi-institutional team. As apheresis blood donation continues to affect more people, the importance of understanding the effects of repeated exposure to citrate on donor skeletal health is essential in protecting this precious community resource.

ELIGIBILITY:
Inclusion Criteria:

* male
* eligible volunteer blood donor
* ≥ 18, and, ≤ 65 years of age at enrollment
* ≥ 1, and, ≤ 5 prior apheresis blood donation procedures

Exclusion Criteria:

* female
* age < 18 or > 65 years at enrollment
* ineligible for whole blood donation
* BMD Z-score <(-2.0) or >(2.0) at any measurement site upon baseline assessment
* metal prosthesis at measurement site
* weight > 300 lbs (136 kg)
* previous fracture of the lumbar spine or femoral neck
* any fragility fracture, defined as a fracture resulting from a fall of standing height or less, during adulthood (specifically ≥18 years of age at the time of fracture)
* previous lumbar spinal fusion surgery
* cystic fibrosis
* emphysema
* celiac disease
* Crohn's disease
* Current or past (>1 month duration) use of medications known to affect BMD including, not limited to: (phenytoin, phenobarbital, corticosteroids)
* Current Osteoporosis Medication use including, but not limited to: (Forteo, oral biphosphonates, Reclast, Prolia, calcitonin)
* Unable or unwilling to donate high frequency apheresis

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Dual Energy XRay Absorptiometry - Total Lumbar Spine | one year
  The primary outcome measure is a decline in total lumbar spine bone mineral density that exceeds the technologist's least significant change (LSC) as assessed by DXA.

SECONDARY OUTCOMES:
Dual Energy XRay Absorptiometry - Femoral Neck | one year
  A secondary outcome measure includes a decline in left or right femoral neck bone mineral density that exceeds the technologist's least significant change (LSC) as assessed by DXA.
Dual Energy XRay Absorptiometry - Total Hip | one year
  A secondary outcome measure includes a decline in total hip bone mineral density that exceeds the technologist's least significant change (LSC) as assessed by DXA.
Dual Energy XRay Absorptiometry - Total Body Composition | one year

CONTACTS AND LOCATIONS:
Overall Officials: Paula E Papanek, PhD, Study Chair — Marquette University; Walter Bialkowski, MS, Study Director — Versiti Blood Health; Robert D Blank, MD, PhD, Principal Investigator — Medical College of Wisconsin; Jerome L Gottschall, MD, Principal Investigator — Versiti Blood Health; Cheng Zheng, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- BloodCenter of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No